CLINICAL TRIAL: NCT02396160
Title: The Effect of Urox™(Crateva, Horsetail and Lindera Combination) in the Treatment of Overactive Bladder and Urinary Incontinence
Brief Title: The Effect of Urox™ in the Treatment of Overactive Bladder and Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: University of Tasmania (Other); Seipel Group Pty Ltd (Industry); Endeavour College of Natural Health (Unknown)
Responsible Party: Principal Investigator, Dr Niikee Schoendorfer, Research Fellow, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SG-04
Record Dates: First submitted 2015-03-17; First posted 2015-03-24 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Overactive Bladder; Urinary Incontinence; Urinary Frequency or Urgency Adverse Event; Nocturia
Keywords: overactive bladder; urinary incontinence; nocturia; urinary frequency
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Nocturia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): 2 capsules per day of the herbal formula (Urox®) with each capsule containing 420mg of a concentrated proprietary blend of extracts of Crateva nurvala stem bark, Equisetum arvense stem and Lindera aggregata root
  Interventions: Dietary Supplement: Urox
- Placebo (Placebo Comparator): identical placebo vegetarian capsule containing color-matched cellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Urox — Active treatment - Proprietary combination of Crateva nurvala, Equisetum arvense and Lindera aggregata herbs
  Arms: Treatment
Other: Placebo — Placebo - Identical vegetarian capsule containing color-matched cellulose to that of the active treatment
  Arms: Placebo

SUMMARY:
This study aims to assess the efficacy of a specialized herbal formula, Urox, versus control over 8 weeks, in a double blind, placebo controlled trial. 150 participants are being recruited, randomized and administered treatment or placebo for the period of 8 weeks after initial eligibility screening. Outcome measures include previously validated tools such as the 3 day symptom diary measuring self-recorded day frequency, nocturia, urgency and incontinence episodes. Quality of life improvements are being measured using the Incontinence Impact Questionnaire, Urinary Distress Inventory and the short version of the OverActive Bladder survey.

DETAILED DESCRIPTION:
Initial consultations were held at either the Brisbane campus of the Endeavour College of Natural Medicine Naturopathic clinic or at Kelvin Grove Natural Medicine clinic, Brisbane. Follow up interviews are being conducted via telephone. To minimize dropout rates, participants are telephoned (as a reminder for the call and to complete the micturition diaries) approximately 1 week before the scheduled interview time and were intermittently called over the week following if they were unable to be reached at the scheduled interview time. Three attending clinicians interviewed trial participants, all having participated in interview training prior to any interviews being taken. The training was designed to ensure utility of a uniform and consistent approach regarding how questions were asked and how data was recorded.

The week prior to an initial consultation participants were requested to complete a micturition diary and health related quality of life surveys, to serve as baseline measures. The attending clinician then also completed a clinical data sheet, at the time of the initial consultation, containing a range of questions including demographics, exercise, health history and habits, which will be used to control and correlate data variables. Any incomplete quality of life surveys at the outset were also completed at the first interview.

Micturition diaries are collected by post at 2, 4 and 8 week intervals along with the completion of quality of life surveys and follow up clinical data sheet via telephone. Participants were asked to keep the micturition diary for 3 days prior to each consultation and were provided reply paid envelopes to return the surveys and unused capsules to assess compliance.

For the primary outcome (day frequency) measure it was calculated that 90 participants equally divided into placebo and control were required to detect a difference of 1.6 urinary frequency episodes per day (2.7SD) between treatment and placebo groups, with a two-tailed alpha of 0.05 and a power of 80%. For total incontinence, 53 participants were required equally divided into each group to detect a difference of 1.2 episodes per day (2.2SD), while for urgency 54 was required in each group to detect a difference of 2 per day (3.7SD). To account for potential drop-outs and variations in presenting symptoms, a total of 150 participants were recruited.

Data for the two treatments will be compared using mixed effects ordered logistic regression adjusted for repeated measures (Stata, version 13.1, StataCorp, TX, USA). GraphPad Prism (version 6.00 for Windows, GraphPad Software, La Jolla California, USA) will be used to plot the data. Data (day frequency, night frequency, urgency and incontinence) will be evaluated by intention to treat analysis, with the last result brought forward for people who dropped out or were lost to follow-up. Variables selected for adjustment using backward stepwise regression from list including age, sex, water intake and diuretic use (p<0.22 for covariate inclusion). Holm estimation test will be used to adjust p-values for repeated measures. Each analysis will only included participants who are symptomatic at baseline. For example, in relation to daytime urinary frequency - only participants with baseline of ≥10 will be included in the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include symptoms of urinary frequency (at least ten times per day) and/or incontinence (at least nine episodes per week), provided they have experienced symptoms of OAB for at least 6 months.

Exclusion Criteria:

1. Recent surgery particularly hysterectomy or prolapse repair (within the last 12 months)
2. Recently undergone childbirth (within the last 12 months), or currently pregnant.
3. Use of any natural therapies for bladder symptoms in the last month.
4. Concomitant health conditions such as uncontrolled diabetes mellitus, heart disease, pancreatic, hepatic or renal disease, recurrent urinary tract infections, and chronic inflammatory conditions, which may otherwise affect outcomes.
5. Currently being treated for mental health issues or psychiatric disturbances.
6. Any individuals who are presently taking prescribed medication for incontinence or OAB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niikee Schoendorfer, PhD, Principal Investigator — The University of Queensland

IPD SHARING:
Plan to Share IPD: No
As data was analysed de-identified, it is not possible to have individual participant data available associated with their name and details.

REFERENCES:
- [Derived] Schoendorfer N, Sharp N, Seipel T, Schauss AG, Ahuja KDK. Urox containing concentrated extracts of Crataeva nurvala stem bark, Equisetum arvense stem and Lindera aggregata root, in the treatment of symptoms of overactive bladder and urinary incontinence: a phase 2, randomised, double-blind placebo controlled trial. BMC Complement Altern Med. 2018 Jan 31;18(1):42. doi: 10.1186/s12906-018-2101-4. PMID 29385990

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 75 | 75
Completed | 69 | 73
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Population: This data includes all those who met criteria (minimum of 2 of the following symptoms per day for 6 months - Urinary Day Frequency ≥10 daytime micturitions; Nocturia ≥2 night time micturitions; Urinary Urgency ≥2 episodes and/or Incontinence ≥1 episode) and were entered into randomisation at the commencement of their enrollment into the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.21 (12.11) | 62.26 (13.87) | 63.23 (13.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 48 | 88
  Male | 35 | 27 | 62
Weight [Mean (Standard Deviation); unit: kg] | 79.90 (18.78) | 79.73 (22.74) | 79.82 (20.81)
Day urinary frequency [Number; unit: participants] — number of participants ≥10 daytime micturitions per day
  participants | 50 | 57 | 107
Night urinary frequency [Number; unit: participants] — number of participants ≥2 nocturnal micturitions per night
  participants | 70 | 61 | 131
Urgency [Number; unit: participants] — number of participants ≥2 urgency micturitions per day
  participants | 62 | 62 | 124
Urge incontinence [Number; unit: participants] — number of participants ≥1 urge incontinent episode per day
  participants | 34 | 35 | 69
Stress incontinence [Number; unit: participants] — number of participants ≥1 stress incontinent episodes per day
  participants | 11 | 10 | 21
Any incontinence [Number; unit: participants] — number of participants ≥1 any incontinence episodes per day
  participants | 35 | 43 | 78
2 symptoms [Number; unit: participants] — number of participants reporting meeting 2 symptom criteria per day
  participants | 24 | 23 | 47
3 symptoms [Number; unit: participants] — number of participants reporting meeting 3 symptom criteria per day
  participants | 33 | 29 | 62
4 symptoms [Number; unit: participants] — number of participants reporting meeting 4 symptom criteria per day
  participants | 18 | 23 | 41

OUTCOME MEASURES:

1. Primary Outcome: Day Urinary Frequency
Description: Day urinary frequency as defined as the number of voluntary diurnal micturitions per day, recorded in a validated urinary diary
Time Frame: 8 weeks
Population: Analysis includes participants who met the criteria for this outcome being day urination frequency ≥10 daytime micturitions per day at baseline. Please note that not all participants in this study met the criteria for all outcomes, hence numbers in each section may seem incongruent with total study participants.
Measure: Mean (95% Confidence Interval); unit: number of diurnal micturitions per day
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 50 | 57
number of diurnal micturitions per day | 7.68 [7.46 to 7.91] | 10.95 [10.70 to 11.20]

2. Secondary Outcome: Urinary Urgency Frequency
Description: Urinary urgency as defined by number of urgency episodes per day recorded in a validated urinary diary
Time Frame: 8 weeks
Population: Analysis includes participants who met the criteria for this outcome being urgency urination frequency ≥1 per day at baseline. Please note that not all participants in this study met the criteria for all outcomes, hence numbers in each section may seem incongruent with total study participants.
Measure: Mean (95% Confidence Interval); unit: number of urgency episodes
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 62 | 62
number of urgency episodes | 1.49 [1.28 to 1.71] | 3.92 [3.65 to 4.19]

3. Secondary Outcome: Urge Incontinence Frequency
Description: Urge incontinence as defined by number of incontinence episodes per day resulting from urinary urgency, recorded in a validated urinary diary
Time Frame: 8 weeks
Population: Analysis includes participants who met the criteria for this outcome being urge incontinent frequency ≥1 per day at baseline. Please note that not all participants in this study met the criteria for all outcomes, hence numbers in each section may seem incongruent with total study participants.
Measure: Mean (95% Confidence Interval); unit: number of urge incontinence episodes
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 34 | 35
number of urge incontinence episodes | 1.21 [0.89 to 1.54] | 2.36 [2.07 to 2.66]

4. Primary Outcome: Nocturia Frequency
Description: Night time urinary frequency as defined as the number of voluntary nocturnal micturition's per day recorded in a validated urinary diary
Time Frame: 8 weeks
Population: Analysis includes participants who met the criteria for this outcome being nocturnal frequency ≥2 per day at baseline. Please note that not all participants in this study met the criteria for all outcomes, hence numbers in each section may seem incongruent with total study participants.
Measure: Mean (95% Confidence Interval); unit: number of nocturnal micturitions
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 70 | 61
number of nocturnal micturitions | 2.16 [2.02 to 2.29] | 3.11 [2.98 to 3.24]

5. Secondary Outcome: Stress Incontinence Frequency
Description: Stress incontinence as defined by number of episodes of incontinence per day related to stress, recorded in a validated urinary diary
Time Frame: 8 weeks
Population: Analysis includes participants who met the criteria for this outcome being stress incontinence frequency ≥1 per day at baseline. Please note that not all participants in this study met the criteria for all outcomes, hence numbers in each section may seem incongruent with total study participants.
Measure: Mean (95% Confidence Interval); unit: Number of stress incontinence episodes
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 11 | 10
Number of stress incontinence episodes | 0.67 [0.47 to 0.86] | 1.6 [1.26 to 1.94]

ADVERSE EVENTS:
Arm/Group | Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/73
Other Adverse Events (participants affected / at risk) | 5/69 | 8/73
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=69) | Placebo (N=73)
Episodes of diarrhea (Gastrointestinal disorders) | 2 | 2
Urinary tract infection (Renal and urinary disorders) | 2 | 1
Headache and worsened asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Worsened memory (Psychiatric disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Facial flushing (General disorders) | 0 | 1
Halitosis (General disorders) | 0 | 1
Worsened arthritic pain (Musculoskeletal and connective tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Limitations of this study include the relatively short duration and lack of long-term follow up. As a phase 2 clinical trial, there was no active comparator and a smaller sample size was also utilized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No